CLINICAL TRIAL: NCT04030494
Title: Study of Validation of the Advanced Blood Pressure Monitor Withings WPM04 for the Detection of Anomalies of Arterial Pressure, Arrhythmia and Valvular Heart Diseases
Brief Title: Validation Study of an Advanced Blood Pressure Monitor
Acronym: TALISMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A02847-48
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation; Hypertension; Valvular Heart Disease
Keywords: blood pressure; Arrhythmias, Cardiac; atrial fibrillation; valvular disease; blood pressure monitors; electrocardiography; Doppler echocardiography; Heart diseases; Cardiovascular diseases
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Heart Valve Diseases; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood pressure (BP) (Other): Group for the validation of blood pressure measurement by the device
  Interventions: Diagnostic Test: BP measurement; Diagnostic Test: VHD detection
- Atrial fibrillation (AF) (Other): Group for the validation of detection of AF by the device
  Interventions: Diagnostic Test: AF detection; Diagnostic Test: VHD detection
- Valvular heart disease (VHD) (Other): Group for the validation of detection of VHD by the device
  Interventions: Diagnostic Test: BP measurement; Diagnostic Test: AF detection; Diagnostic Test: VHD detection

INTERVENTIONS:
Diagnostic Test: BP measurement — sequential BP measurement with Withings WPM04 and sphygmomanometer with dual observer auscultation
  Arms: Blood pressure (BP); Valvular heart disease (VHD)
Diagnostic Test: AF detection — single lead ECG with Withings WPM04 and 12 lead ECG
  Arms: Atrial fibrillation (AF); Valvular heart disease (VHD)
Diagnostic Test: VHD detection — phonocardiogram with digital stethoscope of Withings WPM04 and Doppler echocardiography

SUMMARY:
The proposed clinical study aims to validate the effectiveness of the WPM04 blood pressure monitor developed by Withings as a diagnostic tool for cardiovascular disorders.

The detection of cardiovascular disorders is oriented along three axes, namely the measurement of blood pressure, the identification of rhythm disorders such as atrial fibrillation and the identification of heart murmur indicating valvular heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old,
* Subject who signed the consent form,
* Subject affiliated to a social security scheme or entitled.

Exclusion Criteria:

* Underage subject;
* Subject who refused to participate in the study;
* Subject participating in other research or clinical studies;
* Subject with body mass index greater than 35 kg/m2;
* Subject in linguistic or psychic incapacity to sign an informed consent;
* Subject with congenital cardiomyopathy;
* Subject with aorto-venous fistula;
* Subject with pulmonary pathology that may degrade the quality of the recording;
* Subject presenting a serious pathology compromising the realization of the examinations envisaged in the test;
* Subject with an arm injury incompatible with the use of an armband sphygmomanometer;
* Subject receiving an intravenous perfusion on the left arm;
* Subject with electrical stimulation by pacemaker, implantable cardioverter-defibrillator;
* Subject with prosthetic heart valve;
* Subject under kidney dialysis;
* Hemodynamically unstable subject (acute heart failure or cardiac assistance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
BP precision and accuracy | 1 visit (45 minutes)
  mean error and standard deviation on measurements, and standard deviation on patients (criteria 1 and 2 of ANSI/AAMI/ISO 81060-2:2013) against sphygmomanometer dual observer auscultation
AF and SR classification accuracy | 1 visit (30 minutes)
  sensitivity and specificity of detection of AF and SR from 1-lead ECG against 12-lead ECG
VHD detection accuracy | 1 visit (30 minutes)
  sensitivity and specificity of detection of VHD from phonocardiogram against Doppler echocardiogram

SECONDARY OUTCOMES:
safety evaluation | 1 visit (1 hour)
  frequency of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique AXIUM Centre de cardiologie, Aix-en-Provence, France

IPD SHARING:
Plan to Share IPD: No